CLINICAL TRIAL: NCT05109325
Title: IntERact: Preventing Risky Firearm Behaviors Among Urban Youth Seeking Emergency Department Care
Brief Title: Project IntERact V2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Carter, Associate Professor of Emergency Medicine; Center Director, OVPR Institute of Firearm Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00188022; R01CE003303 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Firearm Violence; Firearm Carriage; Injury Prevention
Keywords: Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care + assessment (No Intervention): Daily assessments (without delivery of intervention components) will be conducted with EUC participants and they will receive a brochure with violence, substance use, and mental health resources.
- IntERact (Experimental): Participants will receive three remotely delivered behavioral therapy sessions (combining motivational interviewing, cognitive behavioral skills training, and care management), with an smartphone APP supporting the therapy and delivering therapeutic content in-between therapy sessions.
  Interventions: Behavioral: IntERact

INTERVENTIONS:
Behavioral: IntERact — The IntERact intervention includes: (1) three remotely delivered Health Coach therapist sessions that integrate behavioral therapy (motivational interviewing [MI] + cognitive behavioral therapy [CBT] and strengths-based care management (CM); as well as, (2) an APP supporting and enhancing the therapist intervention by: (a) conducting automated daily assessments; (b) delivering daily MI/CBT messages tailored by the daily surveys; (c) delivering GPS-enabled alert notifications and immediate one-touch pro-social support; (d) providing access to reminders regarding goals/strengths from the ED session, CBT tools/skills (e.g., infographics, coping strategies, harm reduction strategies), and other psychoeducation (e.g., safe storage); (e) facilitating one-touch contact with pro-social support, including the health coach and others; (f) providing easy linkage to care management resources (web links, phone numbers, contact information).
  Arms: IntERact

SUMMARY:
The present study is evaluating the efficacy of a behavioral intervention to reduce risky firearm carriage among a high risk sample of youth reporting recent firearm carriage and ownership of a smartphone.

DETAILED DESCRIPTION:
Firearms are the leading cause of death for U.S. youth; 60% due to homicide. This study will test the efficacy of a behavioral intervention at reducing risky firearm behaviors among a high-risk community sample of youth (age 16-24) that report past 3-month firearm carriage and smartphone ownership. The behavioral intervention consists of 3 remotely delivered therapy sessions integrating motivational interviewing (MI), cognitive behavioral therapy (CBT), and care management (CM), supported by a smartphone APP that facilitates therapist contact, conducts automated daily assessments, delivers between session tailored therapy content, delivers just-in-time Global Positioning System (GPS)-triggered notifications upon entry into high-risk locations, and aids with utilization of local resources. Recruitment will proceed in two high-risk communities (Flint, Saginaw), including through the main Emergency Departments/trauma centers that are located in both cities. Given elevated rates of firearm violence among socio-disadvantaged youth with disparities in access to community services, the proposed intervention, if found to be efficacious, has the potential for significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Flint or Saginaw Youth between the ages of 16 to 30 reporting past 3-month firearm carriage and ownership of a smartphone, including those seeking care for any reason at Hurley Medical Center or Covenant Medical Center Emergency Department.
* Can provide consent (age: 18-30) or youth assent and parental consent (age: 16-17) for the study.

Exclusion Criteria:

* Incarcerated (i.e., in active policy custody and not able to provide informed consent)
* Presenting to the ED for active suicide ideation or attempt, sexual assault, and/or child abuse
* Unable to provide informed consent due to mental status (e.g., alcohol intoxication, acute psychosis) or medical instability.
* Participants will be excluded if firearm carriage is exclusively for legal work (e.g., police), hunting, or target shooting.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 373 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Risky Firearm Behaviors | Baseline to 3 months and 6 months
  Composite measure used in prior work (Carter 2019). Composite measure uses items from the Tulane University Youth Study and Conflict Tactics Scale capturing frequency and severity of risky firearm-related behaviors (e.g. carriage, threats, use, etc.). (0=Never; 6=20+ Times)

SECONDARY OUTCOMES:
Change in Aggression | Baseline to 3 months and 6 months
  Aggression will be measured at Baseline, 3 months, 6 months. Conflict Tactic Scale measures have been used in prior work and is scored using a summary scale. (0=Never; 6=20+ Times).
Change in Victimization | Baseline to 3 months and 6 months
  Victimization will be measured at Baseline, 3 months, 6 months. Conflict Tactic Scale measures have been used in prior work and is scored using summary scale (0=Never; 6=20+ Times).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Carter, M.D., Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Covenant Medical Center, Saginaw, Michigan

IPD SHARING:
Plan to Share IPD: No